CLINICAL TRIAL: NCT02580266
Title: Blood/Urine Markers for Drug Discovery for Renal Disease in Diabetes
Acronym: DDRD
Status: Withdrawn | Type: Observational
Why Stopped: funding withdrew
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Version-2, 01 Sept 2015
Record Dates: First submitted 2015-10-05; First posted 2015-10-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Complications
Keywords: Kidney; Diabetes
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Diabetic nephropathy (kidney problems caused by diabetes) is a devastating chronic vascular complication of diabetes. New treatments are urgently needed for preventing or slowing down the progression of diabetic kidney disease. Samples of serum/plasma/urine will be obtained from patients with diabetes and different degree of renal impairment.

In this project cells in culture will be treated with plasma or serum or urine; cells extracts or supernatant will be studied to screen for modulation (activation/inhibition) of different cellular pathways using gene array, metabolomic and/or proteomic. Once some cellular pathways have been identified specific analysis will be conducted on the biological material collected to confirm specific "cell signatures" that could represent potential target for treatment.

DETAILED DESCRIPTION:
The aim of the study is to investigate novel putative mechanisms involved in the pathophysiology of kidney disease in diabetic patients.

The investigators will make use of plasma, serum or urine obtained from patients with diabetes.

Cells in culture will be treated with plasma or serum or urine; cells extracts or supernatant will be studied to screen for modulation (activation/inhibition) of different cellular pathways using gene array, metabolomic and/or proteomic. Once some cellular pathways have been identified specific analysis will be conducted on the biological material collected to confirm specific "cell signatures" that could represent potential target for treatment.

The investigators will recruit patients with both type 1 and type 2 diabetes attending our outpatient diabetes clinic at Guys' and St Thomas Hospital. The participant will be informed of the aim of the research and if agreeable in donating blood and urine sample; participants will be asked to sign a written informed consent explaining in simple word the aim of the research, the involvement they should have (blood sample and urine sample collection), the minimal risk to which they will be exposed (venopuncture).

The study will involve one or more blood collections from the arm, for up to 30 mls (6 tea spoons) per year (up to 10 yeas duration), to be collected on up to 2 occasions/ year (minimum time between two collections: 4 weeks), with up to 15ml (3 tea spoon) of blood maximum volume taken per occasion. Urine samples (any amount) might also be collected at any time. Blood and urine collections will take approximately 15 minutes.

This research is low risk. Samples will be stored within the Unit of Metabolic Medicine (Dr Gnudi), King's College London, United Kingdom, and its potential future use will be within the remit of the advancement of science and for the benefit of public domain within academic and/or commercial organisations (e.g. pharmaceutical industry) worldwide.

Any information collected from participants during the course of the research will be kept strictly confidential. Any information leaving the hospital will have the name and address of patient removed so that it can not be recognised by third parties.

The results obtained from this research will likely to be published in a medical journal. The investigators will provide copy of any published results to anybody that may request for it. Participants will not be identified in any report/publication.

ELIGIBILITY:
Inclusion Criteria:

* type 1 and type 2 diabetes

Exclusion Criteria:

* major acute cardio (myocardial infarct, stroke, ec) renal (acute renal failure) events, or severe debilitating disease (e.g. cancer) during the 6 months before the blood/urine collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 and type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Cellular phenotype | 5 years
  Cellular phenotype (gene and protein expression level)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Gnudi, MD, PhD, Principal Investigator — King's College London
Locations (1):
- Unit for Metabolic Medicine, King's College London, London, United Kingdom